CLINICAL TRIAL: NCT06892535
Title: Low-Dose Albumin Infusion for the Prevention of Paracentesis Induced Circulatory Dysfunction (PICD), After Large Volume Paracentesis in Decompensated Cirrhosis of Liver.
Brief Title: Low-dose Albumin Infusion for the Prevention of Paracentesis Induced Circulatory Dysfunction (PICD), After Large Volume Paracentesis (LVP) in Decompensated Cirrhosis Liver.
Acronym: PICD LVP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Abu Md Asaduzzaman, Thesis student of Doctor of Medicine (MD), Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 4794; BSMMU/2024/1784 (Other Grant/Funding Number: BSMMU)
Record Dates: First submitted 2025-03-19; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-02

CONDITIONS: Paracentesis-Induced Circulatory Dysfunction
Keywords: Low dose albumin infusion for PICD prevention after LVP in Decompensated cirrhosis

STUDY DESIGN:
Intervention Model Description: Low dose albumin infusion compared with standard dose albumin infusion after large volume paracentesis in decompensated cirrhosis of liver.
  Intervention group: Low dose albumin. Control group: Standard dose albumin. Randomization was made by using the Random Allocation Software, version 1, 2022.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Albumin infusion, 6gm/L of ascitic fluid aspiration. (Active Comparator)
  Interventions: Drug: Albumin infusion, 2g/L of ascitic fluid aspiration.

INTERVENTIONS:
Drug: Albumin infusion, 2g/L of ascitic fluid aspiration. — Albumin infusion lower than the standard dose, either 2g/L or 4g/L of ascitic fluid aspiration is termed as low dose.

SUMMARY:
Abstract for thesis protocol. Background: Paracentesis induced circulatory dysfunction (PICD) is a common complication of large volume paracentesis in cirrhotic patients, which can lead to renal impairment, hyponatremia, and increased mortality. Albumin infusion is recommended to prevent PICD, but the optimal dose is unclear. We aim to compare the efficacy of low dose albumin infusion versus standard dose of albumin in preventing PICD in cirrhotic patients.

Material and methods: We will conduct a randomized controlled trial with two arms: low dose albumin infusion (2g per liter of ascitic fluid removed) versus standard dose albumin infusion (6g per liter of ascitic fluid removed). Patients with liver cirrhosis undergoing large volume paracentesis (>5 L) with serum creatinine <1.5 mg/dL and no signs of infection will be included in the study.

Sample size calculation: Based on previous studies, group sample size will be 26 and will achieve 80.749% power to reject null hypothesis. As per availability, 30 participants will be included in each group, with a total number of 60 for this trial.

Outcome of the study:

The primary outcome is the incidence of paracentesis induced circulatory dysfunction (PICD) in both groups, (Low dose albumin and standard dose of albumin), 7 days after paracentesis.

The secondary outcomes are renal failure, hyponatremia, hepatic encephalopathy, hepatorenal syndrome, and length of hospital stay.

Conclusion: This trial will provide evidence on whether low dose albumin infusion is as effective as standard dose albumin infusion in preventing PICD in cirrhotic patients. This could have implications for reducing the cost and optimal effective dose of albumin therapy, as well as improving the outcomes of patients with ascites.

DETAILED DESCRIPTION:
Introduction. Cirrhosis of liver is the almost final pathway of chronic liver disease, leading to hepatocellular carcinoma that become critical when it progress to decompensation, denotes 13th most common cause of death worldwide (Bai et al., 2022; Carvalho & Machado, 2018).

Ascites is the most common sign of decompensation, that markedly increase mortality in 5 years (Carvalho & Machado, 2018). Approximately 20% of patients become diuretic resistant, who were diuretic responders; and among them 10% become refractory, either due to resistance to diuretics or diuretic-intractable, because of contraindication (Alsebaey, A. et al., 2020).

Till now, apart from liver transplantation (LT), trans jugular intrahepatic portosystemic shunt (TIPS) and large volume paracentesis (LVP) are the available option for the treatment of refractory ascites, but due to chances of recurrence and hepatic encephalopathy, as well as unavailability of TIPS in some places, LVP becomes the only preferred option (Alsebaey, A. et al., 2020; Kulkarni et al., 2020; Singh et al., 2023).

Paracentesis induced circulatory dysfunction (PICD), develops invariably after LVP (Alsebaey, A. et al., 2020), leading fall of intra-abdominal pressure, that initiates increased venous return, increased CO, and decreased renin-angiotensin-sympathetic system, if plasma expander is not used (Kulkarni et al., 2020).

If volume expander not infused within 12 hours, renin-angiotensin-sympathetic system markedly activated with reduced CO, resulting in circulatory imbalance, and PICD developed (Sola-Vera et al., 2003).

Also, there is a hypothesis, LVP leading hypotension, that causes increased bacterial translocation, as well as innate immune activation resulting vasodilation, and consequently PICD developed (Sola-Vera et al., 2003).

As we know, albumin has antioxidant, immunomodulatory, and endothelial stabilization effect, as well as possessing increased oncotic pressure (Carvalho & Machado, 2018,). Studies have established the use of human albumin infusion for the prevention of paracentesis-induced circulatory dysfunction (PICD) in patients with liver cirrhosis requiring large volume paracentesis, (Carvalho & Machado, 2018, Gines et al.,1996).

A decade of research, various agents were used, as the alternatives of albumin; and proves the highest efficacy of albumin compared to terlipressin, noradrenaline, midodrine, synthetic colloids and saline preventing PICD (Gines et al., 1996; Moreau et al., 2006).

LVP, paracentesis of ascitic fluid >5L, leading paracentesis induced circulatory dysfunction (PICD) in approximately 80% cases, associated with rapid recurrence of ascites, dilutional hyponatremia, hepatorenal syndrome (HRS), and increased short-term mortality (Alsebaey, A. et al., 2020).

PICD is defined as increase in plasma renin activity by >50% of baseline to an absolute value of >4ng/ml/h at 6th day, after paracentesis, resulting patients develop rapid reaccumulation of ascites, hyponatremia, renal injury, and hepatic encephalopathy. (Singh et al., 2023, Alsebaey, A. et al., 2020).

Patients with ascites usually have hypoalbuminaemia. Combination of hypoalbuminaemia and impaired albumin function leads to marked disturbance in the transport, metabolism, and excretion of many endogenous and exogenous substances, whereas infusion of exogenous albumin serves the dual purpose of replenishing the level of circulating albumin and the functional activity of albumin pool (Kulkarni et al., 2020).

Volume expansion with albumin infusion is the mainstay of treatment. The use of vasoconstrictors can also help in treatment but needs to be evaluated. Nevertheless, avoiding paracentesis and withholding diuretics and/or betablockers during PICD presents the worsening of hemodynamics and encephalopathy (Kulkarni et al., 2020).

Very few studies have compared low-dose albumin infusion (2 g/L or 4g/L of ascitic fluid removed) with standard-dose albumin (6g-8g/L of ascitic fluid removed) for the prevention of PICD in LVP (Alsebaey, A. et al., 2020, Alessandria et al.,2011).

This study aims to re-evaluate efficacy of low dose albumin infusion (2g/L) compared to standard dose (6g-8g/L of ascitic fluid paracentesis) for the preventing PICD, that might certainly reduce the treatment cost as well as exploring the effectiveness of low dose albumin infusion in this regard, which would be new insight for the future research in management.

LVP results in mechanical decompression of the splanchnic vascular bed, leading vasodilation, a further decrease in the arterial filling, and activation of neurohormonal systems, that causes free water and sodium retention. Consequently, patients develop rapid reaccumulation of ascites, hyponatremia, renal injury, and hepatic encephalopathy (Kulkarni, A.,2020).

Maintaining the intraabdominal pressure by pneumatic girdle prevents circulatory disturbance resulting after paracentesis (Kulkarni, A.,2020).

Peritoneo-venous shunt proponents that ascites will have unidirectional flow from abdomen into the systemic circulation, leading to expansion of effective arterial blood volume, increase in cardiac output (CO), renal blood flow, right atrial pressure, and atrial natriuretic peptide concentration and decrease in renin aldosterone concentrations. As there are arguments and complications, including sepsis, coagulopathies, and pulmonary edema this procedure has not been accepted widely (Kulkarni, A.,2020).

The degree of activation of renin-angiotensin-aldosterone system and sympathetic nervous system 6 days after paracentesis correlates inversely, with changes in systemic vascular resistance (SVR). Within 60 minutes of paracentesis (>5 L), a marked increase in cardiac output (CO), together with a reduction in mean arterial pressure (MAP), and consequently calculated SVR significantly decreased (Kulkarni, A.,2020., Sola-Vera et al., 2003).

Also, there is an increased CO and plasma renin activity (PRA), together with decreased central venous and wedge pressure 24 hours after LVP, and the rate of paracentesis does not have impact on development of PICD; and also study showed, all patients having LVP, have lowered creatinine clearance from 77 to 60 ml/min after 48 hours, irrespective of whether they are edematous or not (Lijnen, et al.,1981).

Rationale of study.

The use of human albumin infusion for the prevention of paracentesis-induced circulatory dysfunction (PICD) in patients with liver cirrhosis requiring large volume paracentesis. A decade of research shows, various agents were used as the alternatives of albumin; but albumin proves the highest efficacy compared to terlipressin, noradrenaline, midodrine, synthetic colloids and saline preventing PICD.

Several studies recommended 6-8g of albumin infusion for each liter of ascitic fluid removal. But the effective dose of it remains elusive still now. Albumin is not only a simple plasma expander, but also possesses antioxidants, immunomodulatory, endothelial stabilization, and platelet antiaggregating effect. Albumin exerts 75% of colloidal osmotic pressure that maintain effective plasma volume. Albumin is associated with high treatment cost; hence, it is warranted to evaluate its efficacy preventing PICD, with lowest possible dose.

Very few studies have compared low-dose albumin infusion (2g/L or 4g/L of ascitic fluid removed) with standard-dose albumin (6g-8g/L of ascitic fluid removed) for the prevention of PICD in LVP.

This study aims to re-evaluate efficacy of low dose albumin (2g/liter of ascitic fluid paracentesis) compared to standard dose (6g-8g/ liter ascites fluid paracentesis) preventing PICD, that might certainly reduce the treatment cost as well as exploring the effectiveness of low dose albumin infusion in this regard, which would be a new insight for future research in the plan of low cost management of decompensated cirrhosis of liver in Bangladesh as well as global perspective.

Research question:

Is there any difference in the outcome between low dose albumin and standard dose albumin infusion, preventing paracentesis induced circulatory dysfunction (PICD), after large volume paracentesis (LVP)?

Literature review:

As we know, in case of refractory ascites in liver cirrhosis large volume paracentesis is warranted to dry up ascites, but risk of developing PICD a dangerous consequence, for which albumin infusion is recommended 6-8 g per liter of ascitic fluid aspiration (Singh et al., 2023).

Alessandria et al., 2011, for the first time infused 4 gm of albumin for each liter of ascitic fluid aspiration to prevent PICD in liver cirrhosis patients. It was studied by Department of Gastroenterology and Hepatology at San Giovanni Battista Hospital, University of Turin, Italy. In this prospective, unblinded, randomized controlled pilot study, was done over 70 participants.35 of them were given 4 gm of albumin infusion for each liter of ascitic fluid aspiration (group-1), on the other hand, rest 35 were given 8 gm of albumin infusion(group-2) (Alessandria et al., 2011). Results of the study revealed PICD (14% vs 20 in group 1 and group 2 respectively; p=ns), hyponatremia (9% vs 6%, p=ns) and renal impairment (0% in both groups) was same in both groups at the 6th day of paracentesis, and 6 months survival as well as recurrent ascites requiring another LVP were also the same.

The study suggested, half dose albumin infusion in cirrhosis patients requiring LVP, effectively prevent PICD and related complications(Alessandria et al., 2011).

Alsebaey, A. et al, in 2020, studied the efficacy of low-dose albumin infusion to prevent PICD and related morbidity, particularly, those who had liver cirrhosis needed LVP. The study was conducted by department of Hepatology and Gastroenterology, National Liver Institute, Menoufia University, Egypt. Total participant of the study was 110, of which 85 participant received low dose albumin (2 gm/L ascitic fluid removed) compared with 25 participant received standard dose albumin infusion (6gm/L ascitic fluid removed).

The study suggested low-dose albumin infusion in cirrhosis patients requiring LVP, was comparable in effective prevention of PICD and related complications (Alsebaey et al., 2020), which supported the study of Alessandria et al., 2011.

In 2022, Bai et al., conducted a systematic review and meta-analysis of multicentered, multinational retrospective RCT of 42 study, of whom, 12 RCT's from Spain,6 in Italy,5 in India, 4 in France, 3 in Egypt, 2 in UK, 2 in China, in Mexico, 2 in Germany and I study from each of the country, Argentina, USA, Iran, and Pakistan. In this study, among the 1608 participant of liver cirrhosis requiring LVP, human albumin received 806 and showed better outcome, and reduced complication related mortality compare with control (OR=0.67, 95% CI=0.67-0.98, p=0.03); also, significantly reduce short-term mortality (OR=0.67, 95% CI=0.50-0.89, p=0.005).

The study suggests that human albumin improves the outcome of cirrhosis patient, however dose is still elusive.

Tan et al.,2016, had conducted a study of 57 participants (n-57), who had undergone paracentesis not more than 8 liters. In this study standard dose (6g/liter of ascitic fluid removed) of albumin was used to prevent PICD. PICD developed 40.3% with no renal impairment. MAP decreased on day 6 compared to baseline. The result of the study found comparable risk of hospital stay, SBP, and other infections, as well as gastrointestinal bleeding and survival.

Richard Moreau et al.,2006, conducted a study comparing synthetic colloid, 3.5% polygeline over albumin for prevention of PICD, cirrhotic patient requiring LVP. Among total 68 participants (n=68) 30 received albumin, over 38 received polygeline. The study was blinded either 8g albumin or 17.5% g polygeline. Dose of albumin was fixed as

1. U If below 4L
2. U If between 4L and 6 L
3. U If between 6L and below 8L
4. U If between 8L or more

Participants were followed over 6 months and evaluated the outcome and complications. The polygeline group revealed a 1.6-fold increased risk of liver related complications than albumin group.

In 2003, Sola-vera J et al., conducted an RCT comparing saline infusion over albumin infusion preventing PICD in Cirrhosis undergoing LVP. Among the 72 participants (n=72), 35 received 3.5% saline infusion, compared to 37 received 20% human albumin 8 g/l of ascitic fluid tap. In this study 10 participants had complications in saline group compared to 6 in albumin group. Incidence of PICD in saline group as 33.3%, compared to 11.4% in albumin group. The study suggested albumin infusion significantly reduced the PICD in liver cirrhosis requiring LVP.

In 1988, Pere Gines conducted a study of 105 participants with liver cirrhosis requiring LVP. Among them 52 received albumin 40g with each tap, compared with no volume expander in other group. Acute kidney injury (AKI) and hyponatremia significantly higher with the participant who had not receive albumin infusion.

In 1996, Gines et al., conducted an RCT, evaluated the efficacy of albumin over dextran 70 and polygeline for the prevention of PICD. In this study, 289 participants undergoing LVP and found in albumin group, PICD was significantly reduced (18.5%), compared to 34.4% in dextran 70 and 37.8% in the polygeline group.

Objectives of the study:

The general objective. To observe and compare the incidence of paracentesis induced circulatory dysfunction (PICD) with low dose albumin and standard dose of albumin, 7 days after large volume paracentesis.

The specific objectives are. To observe and compare the development of complications, including renal failure, hyponatremia, hepatic encephalopathy, and hepatorenal syndrome in both groups after large volume paracentesis.

To observe and compare the length of hospital stay in both groups after large volume paracentesis.

Materials and Methods. We will conduct a randomized control trial comparing low dose albumin infusion (2g per liter of ascitic fluid removal) with standard dose albumin infusion (6g per liter of ascitic fluid removal) preventing paracentesis induced circulatory dysfunction (PICD).

Sampling Technique: Randomized sampling who meet the inclusion criteria. Sample Size Calculation: Alternate Hypothesis π1≠ π0 Here, ((u+v)²(α1²+α0²))/(π1-π_0 )² u= 1.96 v= 0.84 π1=9.0 (π1, mean Plasma renin activity at 6th day, Alessandria et al.,2011) π0=9.8 (π0, mean Plasma renin activity at day "0", Alessandria et al.,2011) α0=1, α1=1 Group sample sizes of 26, and 26 achieve 80.749% power to reject null hypothesis of equal means when the population mean difference is π0-π=9.8-9.0=0.8 with standard deviations of 1.0 for group-1 and 1.0 for group-2, and with a significance level (alpha) of 0.0500 using two-sided two-sample unequal-variance t-test.

As availability, we plan to include 30 participants in each group, with a total number of 60 for this trial.

Selection of participants.

1. Inclusion criteria:

   1. Cirrhotic patients with grade-III ascites.
   2. Age 18 to 80 years.
   3. Willing to consent for clinical trial.
2. Exclusion criteria:

   1. Acute liver failure.
   2. Impaired consciousness.
   3. Patients with following concomitant diseases,

      1. Severe cardiac diseases, respiratory diseases, and Renal impairment, (S. Creatinine >1.5 mg/dl).
      2. Hyponatremia.
      3. Advanced HCC (>3 nodule, portal vein thrombosis)
      4. Hepatic encephalopathy,
      5. Sepsis,
      6. Recent bleeding, e.g., GIT hemorrhage within 7 days before study.
      7. Pregnancy.
   4. Unable or not willing to consent for clinical trial.

Outcome of the study:

1. The primary outcome is the incidence of PICD in both groups (low dose albumin and standard dose albumin), 7 days after paracentesis.
2. The secondary outcomes are renal failure, hyponatremia, hepatic encephalopathy, development of hepatorenal syndrome, length of hospital stay, and mortality.

   Study design.

   Type of Study: Randomized Control trial. Study Period: From IRB clearance to February 2025. Place of Study: Department of Hepatology, Bangabandhu Sheikh Mujib Medical University, Dhaka.

   Study Population: Liver cirrhosis patient with grade-III, ascites requiring large volume paracentesis, (LVP).

   Material and methods: We will conduct a randomized controlled trial comparing the efficacy of low dose albumin infusion (2g per liter of ascitic fluid removal) with standard dose albumin infusion (6g per liter of ascitic fluid removal) preventing paracentesis induced circulatory dysfunction (PICD) in decompensated cirrhosis of liver.

   Randomization procedure: Randomization will be made by using the Random Allocation Software, version 1, 2022.

   Study procedure. Participants who meet the inclusion criteria will be taken. All participants will be on a low salt diet and without diuretic therapy at least 3 days prior paracentesis. On the day '0' primary assessment will be performed with body weight, mean arterial pressure (MAP), heart rate, complete blood count (CBC), Prothrombin time (PT), International normalization ration (INR), liver function test, (Serum Bilirubin, Serum Alanine aminotransferase, ALT, Serum Aspartate aminotransferase, AST, Serum Albumin), renal function test (serum creatinine & electrolyte), and Plasma renin activity (PRA).

   Blood samples will be taken after an overnight fast and bed rest for at least 30 minutes in supine position, for measuring PRA. Samples will be sent to the laboratory in EDTA labeled vacuum tube (lavender blood tube) and centrifuge at 2500 rpm for 10 minutes and will be stored at '-20' degree centigrade.

   Paracentesis (>5L) will be done with aseptic precautions. Patient should be on lateral decubitus position with empty bladder. An injection needle of 20-22 gauge, or routine blood transfusion set is usually used. The needle is to be inserted as Z-track method on iliac region at the point of distal 2/3rd to the meeting line of umbilicus and anterior superior iliac spine. Paracentesis fluid is to be collected in a plastic bag or container. After paracentesis, bandage is to be applied with sterile gauge. Patient is to be advised not to lie on the paracentesis site. After 24 hours the bandage is to be removed.

   All participants will receive 20% Human albumin, of which 50% of dose within 1 hour of paracentesis. Patients will be treated with albumin in two groups, which will be selected randomly; Intervention group will get 2g, albumin whereas control group will get 6g, per liter of ascitic fluid paracentesis. Randomization will be made by using the Random Allocation Software, version 1, 2022.

   On day 6, blood samples will be taken for Complete blood count (CBC), Prothrombin time (PT), International normalization ratio (INR), Bilirubin, Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), Albumin, Creatinine, Electrolyte, Plasma renin activity (PRA). Changes in effective arterial blood volume will be evaluated, measuring PRA.

   Biochemical and Laboratory Analysis:

   All laboratory tests, Complete blood count (CBC), Prothrombin time (PT), International normalization ratio (INR), Bilirubin, Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), Albumin, Creatinine, Electrolyte, Plasma renin activity (PRA), Ascitic fluid cytology and HBsAg will be done in the department of Laboratory Medicine, Virology, and department of Biochemistry & Molecular Biology, Bangabandhu Sheikh Mujib Medical University, and Ibn Sina trust, Dhaka.

   Data collection technique:

   Following IRB approval, subjects who meet the inclusion criteria, presenting to hepatology inpatient wards at Bangabandhu Sheikh Mujib Medical University, will be approached for participation in the study. Consent will be obtained from the patient or the legally authorized representative if the patient is unable to consent. After consent is signed, the rest of the data will be collected. Medical records will be reviewed in detail during the hospitalization.

   Data analysis plan:

   Data will be analyzed using IBM*, SPSS* Statistics*, version 29 for windows. Data will be expressed mean, ± standard deviation (SD) for nonparametric data, whereas number with column, percentage for nominal data, and range for nonparametric data. All p-values <0.05 will be considered significant. A comparison between 2 groups will be made, using the students' 't' test for parametric data, whereas Mann-Whitney test for nonparametric data.

   Comparison of variables, treatment induced change in the same group, paired 't' test, whereas Wilcoxon signed rank test for nonparametric data.

   Univariate and multivariate binary logistic regression will be done for detecting the predictors of PICD.

   Ethical Consideration.

   Ethical clearance will be taken from IRB, Bangabandhu Sheikh Mujib Medical University, before starting this study. Informed written consent (English/Bengali version) will be taken from each patient. The purpose and procedures will be briefly explained to all participants. The final database and report will not contain the names of participants.

   Use of drugs:

   20% Human albumin, 2g/ liter of ascitic fluid aspiration will be compared with standard dose (6g) in this study.

   Use of hospital records:

   Hospital records, especially the investigation reports, will be needed to fill up the data collection sheet. The data collection sheet will be filled up after taking a brief interview of 20 - 30 minutes from the participants.

   Risk Reduction & data protection. All study data will be stored without identifiers in a secure (locked) location and only authorized study personnel will have access to study records. Only de-identified data will be sent for combined analysis.

   Monitoring & Reporting of Adverse Events. This is a prospective clinical trial. Subjects will receive 20% Human Albumin infusion, under a standard treatment regimen, for which very minimum chances of adverse effect, including allergic reaction, nausea, vomiting, fever and chills, vascular overload, hemodilution and pulmonary edema. Even though, any medical condition as part of this study will be considered adverse or serious adverse events.

   Subject to any Compensation:

   Participants will not be paid for their participation in the study.

   Operational definitions.

   Paracentesis induced circulatory dysfunction (PICD):

   Paracentesis induced circulatory dysfunction (PICD), is defined as an "increase in plasma renin activity by >50% to an absolute value of >4 ng/ml/hr. at day 6 after paracentesis"(Alsebaey,A. et al., 2020; Singh et al., 2023).

   Low dose albumin:

   Albumin infusion lower than the standard dose, either 2g/L or 4g/L of ascitic fluid aspiration is termed as low dose (Alsebaey,A. et al., 2020, Alessandria et al.,2011).

   Standard dose of albumin:

   Infusion of albumin, 6g-8g per liter of ascitic fluid aspiration (Singh et al., 2023, Alsebaey, A. et al., 2020, Alessandria et al.,2011).

   Grade-III, ascites:

   Grade-III or tense ascites is characterized by presence of ascites which is detected clinically with fluid thrill (Singh et al., 2023).

   Large volume paracentesis:

   Removal of >5L of ascitic fluid in one sitting is regarded as large volume paracentesis (Singh et al., 2023).

   Hepatic encephalopathy (HE) The term hepatic encephalopathy (HE) encompasses a wide array of transient and subtle reversible neurologic and psychiatric manifestations usually found in patients with chronic liver disease and portal hypertension, but also seen in patients with acute liver failure. Symptoms may range from mild neurocognitive disturbances to overt coma (Feldman et al. 2015).

   Bacterial peritonitis (SBP):

   The diagnosis of SBP is made when there is a positive ascitic fluid culture and an elevated ascitic fluid absolute PMN count (i.e., at least 250/mm3 [0.25 × 109/L]) without evidence of an intra-abdominal surgically treatable source of infection (Feldman M et al.2015).

   Acute kidney injury (AKI):

   AKI is now defined according to International Club of Ascites, as proposed by the Kidney Disease Improving Global Outcomes (KDIGO) group, as either an absolute increase in serum creatinine of more than or equal to 0.3 mg/dl (≥26.4 μmol/L) in less than 48 h, or by a percentage increase in serum creatinine of more or equal to 50% (1.5-fold from baseline) in less than seven days (Angeli, et al. 2018).

   Hepatorenal syndrome (HRS):

   HRS has been defined as ''a functional renal failure caused by intrarenal vasoconstriction which occurs in patients with end-stage liver disease as well as in patients with acute liver failure or alcoholic hepatitis" (Angeli, P. et al 2018).

   Hyponatremia:

   Hyponatremia develops in approximately 20-30% of cirrhotic patients with ascites and is defined as a serum sodium concentration less than 130 mmol/L.

   References:

   Alessandria, C., Elia, C., Mezzabotta, L., Risso, A., Andrealli, A., Spandre, M., Morgando, A., Marzano, A. and Rizzetto, M., 2011. Prevention of paracentesis-induced circulatory dysfunction in cirrhosis: standard vs half albumin doses. A prospective, randomized, unblinded pilot study. Digestive and Liver Disease, 43(11), pp.881-886.

   Alsebaey, A., Rewisha, E. and Waked, I., 2020. High efficacy of low-dose albumin infusion in the prevention of paracentesis-induced circulatory dysfunction. Egyptian Liver Journal, 10, pp.1-8.

   Bai, Z., Wang, L., Wang, R., Zou, M., Méndez-Sánchez, N., Romeiro, F.G., Cheng, G. and Qi, X., 2022. Use of human albumin infusion in cirrhotic patients: a systematic review and meta-analysis of randomized controlled trials. Hepatology International, 16(6), pp.1468-1483.

   Carvalho, J.R. and Machado, M.V., 2018. New insights about albumin and liver disease. Annals of hepatology, 17(4), pp.547-560.

   Ginés, A., Fernandez-Esparrach, G., Monescillo, A., Vila, C., Domenech, E., Abecasis, R., Angeli, P., Ruiz-del-Arbol, L., Planas, R., Sola, R. and Ginès, P., 1996. Randomized trial comparing albumin, dextran 70, and polygeline in cirrhotic patients with ascites treated by paracentesis. Gastroenterology, 111(4), pp.1002-1010.

   Ginès, P., Titó, L., Arroyo, V., Planas, R., Panés, J., Viver, J., Torres, M., Humbert, P., Rimola, A., Llach, J. and Badalamenti, S., 1988. Randomized comparative study of therapeutic paracentesis with and without intravenous albumin in cirrhosis. Gastroenterology, 94(6), pp.1493-1502.

   Kulkarni, A.V., Kumar, P., Sharma, M., Sowmya, T.R., Talukdar, R., Rao, P.N. and Reddy, D.N., 2020. Pathophysiology and prevention of paracentesis-induced circulatory dysfunction: a concise review. Journal of clinical and translational hepatology, 8(1), p.42.

   Lijnen, P., Fagard, R., Staessen, J. and Amery, A., 1981. Effect of chronic diuretic treatment on the plasma renin-angiotensin-aldosterone system in essential hypertension. British journal of clinical pharmacology, 12(3), pp.387-392.

   Moreau, R., Valla, D.C., Durand-Zaleski, I., Bronowicki, J.P., Durand, F., Chaput, J.C., Dadamessi, I., Silvain, C., Bonny, C., Oberti, F. and Gournay, J., 2006. Comparison of outcome in patients with cirrhosis and ascites following treatment with albumin or a synthetic colloid: a randomised controlled pilot trial. Liver International, 26(1), pp.46-54.

   Singh, V., De, A., Mehtani, R., Angeli, P., Maiwall, R., Satapathy, S., Singal, A.K., Saraya, A., Sharma, B.C., Eapen, C.E. and Rao, P.N., 2023. Asia-Pacific association for study of liver guidelines on management of ascites in liver disease. Hepatology International, pp.1-35.

   Sola-Vera, J., Miñana, J., Ricart, E., Planella, M., González, B., Torras, X., Rodríguez, J., Such, J., Pascual, S., Soriano, G. and Pérez-Mateo, M., 2003. Randomized trial comparing albumin and saline in the prevention of paracentesis-induced circulatory dysfunction in cirrhotic patients with ascites. Hepatology, 37(5), pp.1147-1153.

   Tan, H.K., James, P.D. and Wong, F., 2016. Albumin may prevent the morbidity of paracentesis-induced circulatory dysfunction in cirrhosis and refractory ascites: a pilot study. Digestive diseases and sciences, 61, pp.3084-3092.

   Appendix-I DATA COLLECTION SHEET Department of Hepatology BSMMU, Shahbag, Dhaka-1000.

   Title of the study:

   Low-dose albumin infusion for the prevention of paracentesis induced circulatory dysfunction (PICD), after large volume paracentesis (LVP) in decompensated cirrhosis liver.

   1. SL NO: 2. Date:

   Particulars of the patient:
   1. Name of patient
   2. Age
   3. Sex
   4. Religion
   5. Occupation
   6. Address
   7. Phone

   Etiology of cirrhosis HBV/ HCV/ MAFLD/ WILSON/ AIH/ CRYPTOGENIC/ OTHERS Duration of diagnosis Amount of ascitic fluid drawn

   On examination On Admission At 6th Day
   1. Systolic BP (mm of Hg):
   2. Diastolic BP (mm of Hg):
   3. MAP (Mean arterial pressure)
   4. Pulse:
   5. Temperature (F):
   6. Degree of ascites
   7. Sarcopenia /umbilical hernia/Hydrocele

   Degree of Liver Dysfunction On Admission At 6th Day CTP MELD, Na Intervention Albumin infusion Low dose (2g/liter ascitic fluid aspiration) High dose (6g/liter ascitic fluid aspiration)

   Complications On Admission At 6th Day

   PICD

   Refractory Ascites

   Hyponatremia

   AKI

   HRS

   Hepatic encephalopathy

   Length of Hospital stay Days

   Need for ICU admission

   HDU/ WARD

   Mortality

   Investigation reports On Admission At 6th Day
   1. Hb% (g/dl):
   2. WBC, TC (--x109 /L)
   3. Platelet count (--´109 /L)
   4. ESR (mm in1st hour)
   5. Prothrombin Time
   6. INR
   7. Bilirubin
   8. Albumin
   9. AST (U/L)
   10. ALT (U/L)
   11. S. Creatinine

   10.S. Electrolyte

   11. PRA

   12. HBs Ag:

   13. Anti HCV

   Signature of Data Collector:

   Appendix-II INFORMED WRITTEN CONSENT

   In native language:

ELIGIBILITY:
1. Inclusion criteria:

   1. Cirrhotic patients with grade-III ascites.
   2. Age 18 to 80 years.
   3. Willing to consent for clinical trial.
2. Exclusion criteria:

   1. Acute liver failure.
   2. Impaired consciousness.
   3. Patients with following concomitant diseases,

      1. Severe cardiac diseases, respiratory diseases, and Renal impairment, (S. Creatinine >1.5 mg/dl).
      2. Hyponatremia.
      3. Advanced HCC (>3 nodule, portal vein thrombosis)
      4. Hepatic encephalopathy,
      5. Sepsis,
      6. Recent bleeding, e.g., GIT hemorrhage within 7 days before study.
      7. Pregnancy.
   4. Unable or not willing to consent for clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
The primary outcome | 6th day
  The primary outcome is the incidence of PICD in both groups (low dose albumin and standard dose albumin), 7 days after paracentesis.

SECONDARY OUTCOMES:
The secondary outcomes | 6th day
  The secondary outcomes are renal failure, hyponatremia, hepatic encephalopathy, development of hepatorenal syndrome, length of hospital stay, and mortality.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hepatology, Bangabandhu Sheikh Mujib Medical University. Dhaka, Bangladesh., Dhaka, Shahbag, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided
I could share IPD with the permission of my supervisor, and officials of the University, as we are promised not to share personal data to third party.

REFERENCES:
- [Background] Tan HK, James PD, Wong F. Albumin May Prevent the Morbidity of Paracentesis-Induced Circulatory Dysfunction in Cirrhosis and Refractory Ascites: A Pilot Study. Dig Dis Sci. 2016 Oct;61(10):3084-3092. doi: 10.1007/s10620-016-4140-3. Epub 2016 Apr 5. PMID 27048451
- [Background] Sola-Vera J, Minana J, Ricart E, Planella M, Gonzalez B, Torras X, Rodriguez J, Such J, Pascual S, Soriano G, Perez-Mateo M, Guarner C. Randomized trial comparing albumin and saline in the prevention of paracentesis-induced circulatory dysfunction in cirrhotic patients with ascites. Hepatology. 2003 May;37(5):1147-53. doi: 10.1053/jhep.2003.50169. PMID 12717396
- [Background] Singh V, De A, Mehtani R, Angeli P, Maiwall R, Satapathy S, Singal AK, Saraya A, Sharma BC, Eapen CE, Rao PN, Shukla A, Shalimar, Choudhary NS, Alcantara-Payawal D, Arora V, Aithal G, Kulkarni A, Roy A, Shrestha A, Mamun Al Mahtab, Niriella MA, Siam TS, Zhang CQ, Huei LG, Yu ML, Roberts SK, Peng CY, Chen T, George J, Wong V, Yilmaz Y, Treeprasertsuk S, Kurniawan J, Kim SU, Younossi ZM, Sarin SK. Asia-Pacific association for study of liver guidelines on management of ascites in liver disease. Hepatol Int. 2023 Aug;17(4):792-826. doi: 10.1007/s12072-023-10536-7. Epub 2023 May 26. No abstract available. PMID 37237088
- [Background] Moreau R, Valla DC, Durand-Zaleski I, Bronowicki JP, Durand F, Chaput JC, Dadamessi I, Silvain C, Bonny C, Oberti F, Gournay J, Lebrec D, Grouin JM, Guemas E, Golly D, Padrazzi B, Tellier Z. Comparison of outcome in patients with cirrhosis and ascites following treatment with albumin or a synthetic colloid: a randomised controlled pilot trail. Liver Int. 2006 Feb;26(1):46-54. doi: 10.1111/j.1478-3231.2005.01188.x. PMID 16420509
- [Background] Lijnen P, Fagard R, Staessen J, Amery A. Effect of chronic diuretic treatment on the plasma renin-angiotensin-aldosterone system in essential hypertension. Br J Clin Pharmacol. 1981 Sep;12(3):387-92. doi: 10.1111/j.1365-2125.1981.tb01231.x. PMID 7028060
- [Background] Kulkarni AV, Kumar P, Sharma M, Sowmya TR, Talukdar R, Rao PN, Reddy DN. Pathophysiology and Prevention of Paracentesis-induced Circulatory Dysfunction: A Concise Review. J Clin Transl Hepatol. 2020 Mar 28;8(1):42-48. doi: 10.14218/JCTH.2019.00048. Epub 2020 Mar 26. PMID 32274344
- [Background] Gines P, Tito L, Arroyo V, Planas R, Panes J, Viver J, Torres M, Humbert P, Rimola A, Llach J, et al. Randomized comparative study of therapeutic paracentesis with and without intravenous albumin in cirrhosis. Gastroenterology. 1988 Jun;94(6):1493-502. doi: 10.1016/0016-5085(88)90691-9. PMID 3360270
- [Background] Gines A, Fernandez-Esparrach G, Monescillo A, Vila C, Domenech E, Abecasis R, Angeli P, Ruiz-Del-Arbol L, Planas R, Sola R, Gines P, Terg R, Inglada L, Vaque P, Salerno F, Vargas V, Clemente G, Quer JC, Jimenez W, Arroyo V, Rodes J. Randomized trial comparing albumin, dextran 70, and polygeline in cirrhotic patients with ascites treated by paracentesis. Gastroenterology. 1996 Oct;111(4):1002-10. doi: 10.1016/s0016-5085(96)70068-9. PMID 8831595
- [Background] Carvalho JR, Verdelho Machado M. New Insights About Albumin and Liver Disease. Ann Hepatol. 2018 July - August ,;17(4):547-560. doi: 10.5604/01.3001.0012.0916. PMID 29893696
- [Background] Bai Z, Wang L, Wang R, Zou M, Mendez-Sanchez N, Romeiro FG, Cheng G, Qi X. Use of human albumin infusion in cirrhotic patients: a systematic review and meta-analysis of randomized controlled trials. Hepatol Int. 2022 Dec;16(6):1468-1483. doi: 10.1007/s12072-022-10374-z. Epub 2022 Sep 1. PMID 36048318
- [Background] Alessandria C, Elia C, Mezzabotta L, Risso A, Andrealli A, Spandre M, Morgando A, Marzano A, Rizzetto M. Prevention of paracentesis-induced circulatory dysfunction in cirrhosis: standard vs half albumin doses. A prospective, randomized, unblinded pilot study. Dig Liver Dis. 2011 Nov;43(11):881-6. doi: 10.1016/j.dld.2011.06.001. Epub 2011 Jul 8. PMID 21741331